CLINICAL TRIAL: NCT05809778
Title: Oral Lesions in Patients Dealing With Eating Disorders: an Epidemiological Study
Brief Title: Oral Lesions in Patients With Eating Disorders
Status: Recruiting | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 18/21
Record Dates: First submitted 2023-03-29; First posted 2023-04-12 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Eating Disorders
Keywords: Eating disorders; Pral lesions; Prevention; Prevalence
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Eating disorders (ED) are common among young. Anorexia (AN) and bulimia (BN) are the most prevalent ED. The American Psychiatric Association's guidelines state a 0.3% AN prevalence among young girls and a 0.1 to 4.2% BN prevalence. Men are not excluded: even if ED are more frequent in females (14-18 years), 1 man off to 10 can be diagnosed with ED. Unfortunately, the onset age is decreasing. In the last few years, always more preteens patients are diagnosed with ED: they generally refer a garbled self perception of body image. ED can have oral manifestations, such as: mucosal lesions, dental erosion, glandular hypertrophy, xerostomia and salivary disorders, dental caries These are the most common manifestations observed in patients with eating disorders, after a routine dental visit. There is not strong evidence that dental caries may be directly related to disordered eating habits; as a matter of fact results are controversial. Despite that, all the studies examined agree on the association between signs listed above and food disorders. Univocal percentages have not been reported in the scientific literature. For instance, a systematic review, dated 2016, showed that dental erosion is diagnosed in 45% of ED people, while other studies documented 70% patients affected by erosion. Another example reported is teeth hypersensitivity. According to some studies, 56% of ED patients reported such complaints, instead of other researches documenting 22% hypersensitivity impairment. As for dental caries, results are dissimilar. Authors showed 78% ED subjects diagnosed with dental caries. Other studies reported almost 50% patients with tooth decay, without statistically significant difference in the values between ED people and controls. All these differences are probably due to the different stages of eating disorders and diagnosis, and oral signs found. Different ages are also considered. The primary aim of the study is to evaluate the prevalence of oral cavity lesions among people affected by eating disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of ED
2. Age between 10 and 18 years

Exclusion Criteria:

1. Parents or caregivers not understanding the Italian language
2. Patients affected by other systemic diseases

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients affected by eating disorders
Sampling Method: Non-Probability Sample
Enrollment: 81 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of oral lesions in ED affected patients | At baseline (day 1)
  Mucosal lesions, dental erosion, glandular hypertrophy, xerostomia or other salivary disorders, and dental caries will be examined.

SECONDARY OUTCOMES:
To evaluate the association between presence of oral lesions and type of ED | At baseline (day 1)
  Clinical data will be collected by clinical records
To evaluate the association between presence of oral lesions and patients' global functioning index | At baseline (day 1)
  Patients' global functioning index will be defined by the Global Assessment of Functioning (GAF), an integral part of the standard multiaxial psychiatric diagnostic system. The purpose of including the GAF in DSM-IV as a tool for axis V assessment is to enable clinicians to obtain information about global functioning to supplement existing data about symptoms and diagnoses and to help predict the allocation and outcomes of mental health treatment. The GAF provides a score from 1 to 100: 1 for situation with low functioning; 100 for situation of complete wellbeing.
To evaluate the association between presence of oral lesions and patients' self-perception about oral health | At baseline (day 1)
  Patients' self-perception about oral health will be defined by the Psychosocial Impact of Dental Aesthetics Questionnaire (PIDAQ), evaluating the oral health-related quality of life: 23 items, with a five-point likert scale ranging from 1 to 5 (1 = strongly disagree and 5 = strongly agree), analyzing dental self-confidence, social impact, psychological impact and aesthetic concern. The Italian version was validated in 2014. The possible range of summary scores varied between 0 to 92. Higher scores indicate a greater degree of negative psychosocial impact.

CONTACTS AND LOCATIONS:
Overall Officials: Milena Cadenaro, MD, Study Director — Institute for Maternal and Child Health IRCCS Burlo Garofolo
Locations (1):
- Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste, Trieste, Italy